CLINICAL TRIAL: NCT04293302
Title: Early Postnatal Management of Gestational Brain Sonographic Malformations.
Status: Completed | Type: Observational
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Principal Investigator, Erez Nadir, MD, Senior Neonatologist, Hillel Yaffe Medical Center
Other Study IDs: 0162-19-HYMC
Record Dates: First submitted 2020-02-29; First posted 2020-03-03 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2021-08

CONDITIONS: Brain Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Brain abnormality: Newborn who had any gestational brain sonographic abnormality
  Interventions: Other: No intervention
- No brain abnormality: Newborn who did not have any gestational brain sonographic abnormality
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Gestational sonographic follow up may find some brain malformations. The trial is about to characterize these findings and correlate with the immediate postnatal findings.

DETAILED DESCRIPTION:
Gestational sonographic follow up may find some brain malformations (such as ventricular enlargement, agenesis of corpus callosum, etc.).The trial is about to characterize these findings and correlate with the immediate postnatal findings.

ELIGIBILITY:
Inclusion Criteria:

* All term newborn infants who underwent a neurologic consultation or brain ultrasound.

Exclusion Criteria:

* Prematurity

Max Age: 1 Week | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All infants who were born in Hillel Yaffe medical center during 2010-2019
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Any postnatal clinical neurologic or sonographic brain abnormality | 10 years
  Post natal sonographic brain abnormality or clinical neurologic abnormality

CONTACTS AND LOCATIONS:
Overall Officials: Erez Nadir, MD, Study Chair — Hillel Yaffe Medical Center
Locations (1):
- Neonatal intensive care unit, Hillel Yaffe medical center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghi T, Carletti A, Contro E, Cera E, Falco P, Tagliavini G, Michelacci L, Tani G, Youssef A, Bonasoni P, Rizzo N, Pelusi G, Pilu G. Prenatal diagnosis and outcome of partial agenesis and hypoplasia of the corpus callosum. Ultrasound Obstet Gynecol. 2010 Jan;35(1):35-41. doi: 10.1002/uog.7489. PMID 20020466